CLINICAL TRIAL: NCT04353713
Title: Oral Dextrose Gel to Prevent Early Hypoglycaemia in Very Preterm Infants
Brief Title: Gel for Early Hypoglycaemia Prevention in Preterm Infants
Acronym: GEHPPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0062019
Record Dates: First submitted 2019-12-16; First posted 2020-04-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hypoglycemia in Newborn Infants
Keywords: Prematurity; oral dextrose gel; randomized controlled trial; placebo
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This will be a randomised, double-blinded (using masking), placebo controlled clinical trial. It will involve multiple study sites.
  The study population will consist of infants born at ≤32 weeks gestation. These may include singleton or multiples births.
  Randomisation will be stratified into two groups using gestational age at birth:
  ≤29 weeks
  29+1 to ≤32 weeks
  Randomisation will also be stratified by multi-centre site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention in this study will consist of oral administration of either Dextrose 40% gel or placebo (2% carboxymethylcellulose) gel immediately after stabilisation of the preterm infant in the delivery room.These intervention products will be identically labelled pre-filled syringes. No person involved in either the trial or clinical care of the newborn will ever know the identity of whether dextrose gel or placebo was ever administered to the newborn.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose Gel (Experimental): Dextrose 40% gel will be given immediately following stabilization at birth via massage into the buccal membrane. This will be prior to transport from the Delivery Room to the Neonatal Unit.
  A dose of 1 ml of gel (Dextrose) will be administered to infants born greater than or equal to 29+1 weeks gestation. Prior to administration, a single brief oral suction will be given if required.
  Half the dose of gel (0.5 ml) will be squeezed onto the gloved finger of a person. This half dose will be given on one side of mouth. The remaining half dose (0.5 ml) of gel will be administered to the other side of the mouth.
  A total dose of 0.5 ml of gel (Dextrose) will be administered to infants born less than or equal to 29+0 weeks gestation.
  Half the dose of gel (0.25 ml) will be squeezed onto the gloved finger of administering person. This half dose will be given on one side of mouth. The remaining half dose (0.25 ml) of gel will be administered to the other side of the mouth.
  Interventions: Dietary Supplement: 40% Dextrose Gel
- Placebo (Placebo Comparator): 2% carboxymethylcellulose gel will be given following stabilization at birth via buccal route. This will be prior to in-house transport from the Delivery Room to the Neonatal Unit.
  A standard total dose of 1 ml of placebo gel will be administered to infants born greater than or equal to 29+1 weeks gestation. Prior to administration, a single brief oral suction will be given if required.
  Half the dose of gel (0.5 ml) will be squeezed onto the gloved finger of person. This half dose will be given on one side of mouth. The remaining half dose (0.5 ml) of gel will be administered to the other side of the mouth.
  A total dose of 0.5 ml of gel (Placebo) will be administered to infants born less than or equal to 29+0 weeks gestation.
  Half the dose of gel (0.25 ml) will be squeezed onto the gloved finger of a person. This half dose will be given on one side of mouth. The remaining half dose (0.25 ml) of gel will be administered to the other side of the mouth.
  Interventions: Dietary Supplement: 2% carboxymethylcellulose gel

INTERVENTIONS:
Dietary Supplement: 40% Dextrose Gel — Prophylactic administration of 40% dextrose gel via buccal mucosa to prevent newborn hypoglycemia
  Arms: Dextrose Gel
Dietary Supplement: 2% carboxymethylcellulose gel — placebo
  Arms: Placebo

SUMMARY:
The GEHPPI study is a multicentre placebo controlled randomized controlled trial that aims to prevent early hypoglycaemia in preterm newborns born at ≤32 week's gestation. To do this we will prophylactically administer to these newborns either a small amount of dextrose 40% gel early as possible after birth via the buccal route in the delivery room or a placebo. We hope this dextrose gel will prevent hypoglycemia occurring during the time period needed for the newborns to be transported to the neonatal unit where they will have their venous access inserted.

This trial aims to demonstrate that administering dextrose gel via the buccal route is a simple and rapid method of preventing early hypoglycaemia in this vulnerable patient group.

This trial aims to show that giving dextrose gel via the buccal route is simple and feasible in this premature population.

This trial aims to reduce the need for rescue intravenous dextrose (2ml/kg dextrose 10%) in those babies who are hypoglycaemic at the time of obtaining intravenous access.

DETAILED DESCRIPTION:
Fetal glucose homeostasis in-utero has some very important characteristics: Kalhan et al. showed that from 20 weeks gestation onwards the lower limit for in-utero (foetal) glucose was 3 mmol/L over most of their remaining gestation (Kalhan et al., 1979); Secondly, foetal glucose control in-utero is completely dependent on maternal plasma glucose control and maternal insulin secretion (Stanley et al., 2015); Lastly, steady state glucose utilization rates in term neonates are 4 to 6 mg/min/kg, however at earlier gestational ages (both foetal and preterm infants) these values are higher 8-9 mg/min/kg (Hay, 2006) indicating that preterm infants need an early and reliable glucose source at birth.

A local retrospective audit in our Level 3 Neonatal Unit (King et al., 2018) reviewed 90 patients who were born in-house ≤ 32 weeks gestation with birth weight ≤1500g over 12months in CWIUH (April 2016 - March 2017). Analysis showed that the first blood gas (at the time of first intravenous insertion) was at median 48mins (IQR 15min) life. Data showed that 30 of 90 patients (33.3%) had hypoglycaemia of <1.8 mmol/L at the time of first intravenous access. This hypoglycaemia is at a level below an operational threshold (level at which to intervene) most commonly accepted internationally.

Recommendations from the Pediatric Endocrine Society (2015) are that for high-risk neonates (without a suspected congenital hypoglycaemia disorder), the goal of treatment is to maintain a plasma glucose concentration >2.8 mmol/L for those aged < 48hrs (grade 2+ evidence) (Thornton et al., 2015). However the American Academy of Pediatrics Committee on Fetus and Newborn advise that if asymptomatic, intravenous treatment of hypoglycaemia is not needed until glucose concentrations are < 1.4 mmol/L (within 4hrs after birth) or <2.0 mmol/L (from 4 to 24 h after birth) (Adamkin, 2011). However if symptomatic and blood glucose <2.2 mmol/L they recommend treating immediately (Adamkin, 2011).

Regarding long-term outcomes, in 2006 Boluyt et al. performed the first systematic review of the evidence for neurodevelopmental impairment following hypoglycaemia in the first week of life. They felt that none of the 18 eligible studies identified provided a valid estimate of the effect of neonatal hypoglycaemia on neurodevelopment. The authors provided recommendations about an optimal study design (Boluyt et al., 2006). In 2018 Shah et al. performed a systematic review and meta-analysis which included neonates born ≥32 weeks gestation who had been screened for hypoglycaemia in the 1st week of life. The authors felt that tests of general development in infancy are unlikely to adequately assess the effects of neonatal hypoglycaemia on brain development, but instead future studies will require longer-term end points at least into mid-childhood, including specific tests of visual-motor and executive function (Shah et al., 2018).

Despite the absence of consensus in the medical literature today, this study's investigators feel that tackling the problem of early hypoglycaemia in these very/extremely premature infants will allow a smoother transition from in-utero (foetal) to postnatal (ex-utero) glucose homeostasis. This may have important long-term neurodevelopmental consequences.

Our study aims to tackle this problem of early hypoglycemia in these vulnerable newborns. To do this we will give these newborns a small amount of 40% dextrose gel as early as possible after birth via the buccal route. They will absorb the gel through the small blood vessels located on the inside of their cheeks & gums and it will enter their bloodstream quickly. We hope this gel will prevent hypoglycemia occurring during the time period needed for the newborns to be transported to the neonatal unit where they will have some form of venous access inserted.

As this research is a trial we want to see if this dextrose gel has this beneficial effect or not. To do this we need to compare the dextrose gel to a non-sugar containing gel (called the "placebo"). The placebo gel will contain simple cellulose ingredient but does not contain sugar and will have no effect on blood glucose. Both gels used in the trial will look identical in appearance and neither the researcher nor the patient (nor parent/s) will know whether they received either the dextrose or the placebo gels. Which gel a newborn receives will be assigned at random, immediately prior to the birth. All newborns will be cared for in the same way according to best standard care.

Newborns will not undergo any additional tests as part of the study. Blood glucose levels will be measured as per standard practice at the time vascular access is obtained. Blood glucose values will be measured on either a blood gas analyzer or laboratory glucose. Patient data collected as part of the study will be pseudo-anonymized/ anonymized and stored safely. Consent for participation can be withdrawn at any time.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of infants born at ≤ 32 weeks gestation. These may include singleton or multiples births.

Exclusion Criteria:

* Any newborn where comfort care (palliative approach) is planned for the care of the newborn following delivery. This will often be due to an antenatally diagnosed lethal and/or major congenital anomaly.

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 534 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of newborns with initial hypoglycemia after birth | 30-60 minutes after birth
  Proportion of newborns with an initial plasma glucose value below the operational threshold (<1.8 mmol/L) (32.4 mg/dl)(measured on blood gas machine or laboratory sample) at a time-point when initial intravascular access is successfully obtained by the clinical team

SECONDARY OUTCOMES:
Proportion of newborns with a hypoglycaemia episode < 2.6mmol/L (46 mg/dl) within first 24hrs after birth | 24 hours after birth
  Any hypoglycemic episode < 2.6 mmol/l (46/mg/dl) within first 24 hours after birth
Proportion of newborns with a hypoglycaemia episode <1.8mmol/L (32.4 mg/dl) within first 24hrs after birth | 24 hours after birth
  Any hypoglycaemia episode <1.8mmol/L (32.4 mg/dl) within first 24hrs after birth
Number of episodes of hypoglycaemia <2.6mmol/L (46 mg/dl) within first 24hrs after birth | 24 hours after birth
  Number of episodes of hypoglycaemia <2.6mmol/L (46 mg/dl) within first 24hrs after birth
Proportion of newborns with a hyperglycaemia episode > 10 mmol/L (180 mg/dl) within first 24hrs after birth | 24 hours after birth
  Proportion of newborns with a hyperglycaemia episode > 10 mmol/L (180 mg/dl) within first 24hrs after birth
Proportion of newborns who received rescue IV dextrose within first 24hrs after birth | 24 hours after birth
  Number of subjects who received rescue IV dextrose (2ml/kg of Dextrose 10%) within first 24hrs after birth
Tolerance of buccal gel in delivery room | 30 minutes after birth
  Tolerance of buccal gel (dextrose/placebo): as defined by small/moderate/large spills from the mouth of the newborn
Incidence of symptomatic hypoglycaemia | 24 hours after birth
  This is defined by a modified Whipples Triad: (1) Presence of characteristic clinical manifestations (tremor, lethargy, coma, seizures) (2) coincident with low plasma glucose concentrations measured accurately with sensitive and precise methods, and (3) that the clinical signs resolve within minutes to hours once normoglycaemia has been re-established.
Proportion of newborns who died within the first 12 hours after birth | 12 hours after birth
  Proportion of newborns who died due to any etiology within the first 12 hours after birth
Proportion of newborns who died after 12 hours following birth but prior to discharge home | 6 months
  Proportion of newborns who died due to any etiology after 12 hours following birth but prior to discharge home or transfer to another hospital
Incidence of early bacterial sepsis and/or meningitis | First 3 days after birth
  Incidence of early bacterial sepsis and/or meningitis. This is defined as a positive bacterial growth in either blood and/or cerebrospinal fluid anytime during first 3 days after birth.
Incidence of necrotising enterocolitis (NEC). | 6 months
  Incidence of NEC prior to discharge home or transfer to another hospital. NEC will be defined at either surgery, at post-mortem, or clinically and radiographically.
Proportion of newborns with severe retinopathy of prematurity requiring treatment. | 6 months
  Proportion of newborns with severe retinopathy of prematurity requiring treatment. with either Bevacizumab (Avastin) and/or laser therapy. This will be prior to discharge home and/or transfer to another hospital.
Proportion of newborns with severe (grade III/IV) intraventricular-germinal matrix hemorrhage (IVH-GMH). | 6 months
  Proportion of newborns with severe (grade III/IV) intraventricular-germinal matrix hemorrhage (IVH-GMH). This will be based upon any cranial ultrasound performed prior to discharge or transfer to another hospital.
Proportion of newborns with periventricular leukomalacia (PVL). | 6 months
  Proportion of newborns with any degree of PVL. This will be based upon any cranial ultrasound performed prior to discharge or transfer to another hospital.

CONTACTS AND LOCATIONS:
Overall Officials: John P Kelleher, MB BCH, Principal Investigator — Coombe Women & Infants University Hospital
Locations (5):
- University Hospital Motol, Prague, Czechia
- Ireland (4):
  - Rotunda Hospital, Dublin
  - The National Maternity Hospital, Dublin
  - Coombe Women & Infants University Hospital, Dublin
  - Galway University Hospital, Galway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Background] Boluyt N, van Kempen A, Offringa M. Neurodevelopment after neonatal hypoglycemia: a systematic review and design of an optimal future study. Pediatrics. 2006 Jun;117(6):2231-43. doi: 10.1542/peds.2005-1919. PMID 16740869
- [Background] Hay WW Jr. Recent observations on the regulation of fetal metabolism by glucose. J Physiol. 2006 Apr 1;572(Pt 1):17-24. doi: 10.1113/jphysiol.2006.105072. Epub 2006 Feb 2. PMID 16455683
- [Background] Kalhan SC, D'Angelo LJ, Savin SM, Adam PA. Glucose production in pregnant women at term gestation. Sources of glucose for human fetus. J Clin Invest. 1979 Mar;63(3):388-94. doi: 10.1172/JCI109314. PMID 429559
- [Background] Shah R, Harding J, Brown J, McKinlay C. Neonatal Glycaemia and Neurodevelopmental Outcomes: A Systematic Review and Meta-Analysis. Neonatology. 2019;115(2):116-126. doi: 10.1159/000492859. Epub 2018 Nov 8. PMID 30408811
- [Background] Stanley CA, Rozance PJ, Thornton PS, De Leon DD, Harris D, Haymond MW, Hussain K, Levitsky LL, Murad MH, Simmons RA, Sperling MA, Weinstein DA, White NH, Wolfsdorf JI. Re-evaluating "transitional neonatal hypoglycemia": mechanism and implications for management. J Pediatr. 2015 Jun;166(6):1520-5.e1. doi: 10.1016/j.jpeds.2015.02.045. Epub 2015 Mar 25. No abstract available. PMID 25819173
- [Background] Thornton PS, Stanley CA, De Leon DD, Harris D, Haymond MW, Hussain K, Levitsky LL, Murad MH, Rozance PJ, Simmons RA, Sperling MA, Weinstein DA, White NH, Wolfsdorf JI; Pediatric Endocrine Society. Recommendations from the Pediatric Endocrine Society for Evaluation and Management of Persistent Hypoglycemia in Neonates, Infants, and Children. J Pediatr. 2015 Aug;167(2):238-45. doi: 10.1016/j.jpeds.2015.03.057. Epub 2015 May 6. No abstract available. PMID 25957977
- [Derived] King G, Sloan J, Duddy P, O'Sullivan A, O Cathain N, Miletin J, Dempsey S, Moore S, Purna JR, McDermott C, Moran M, James J, Letshwiti JB, Tabery K, Kubatova A, Janota J, Kelleher J. Delivery room dextrose gel for preterm hypoglycaemia (the GEHPPI study): a randomised placebo-controlled trial. Arch Dis Child Fetal Neonatal Ed. 2025 Apr 17;110(3):319-325. doi: 10.1136/archdischild-2024-327313. PMID 39515988